CLINICAL TRIAL: NCT02771210
Title: A Randomized, Double-blind, Placebo-controlled Multicenter Study of Subcutaneous Secukinumab to Demonstrate Efficacy in the Treatment of Enthesitis at the Achilles Tendon up to 1 Year in Adult Patients With Active Psoriatic Arthritis (PsA) and Axial Spondyloarthritis (axSpA) (ACHILLES)
Brief Title: Study of Efficacy and Safety of Secukinumab in Psoriatic Arthritis and Axial Spondyloarthritis Patients With Active Enthesitis Including One Achilles Tendon Site
Acronym: ACHILLES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F3301; 2016-000972-91 (EudraCT Number)
Record Dates: First submitted 2016-03-31; First posted 2016-05-13 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Psoriatic Arthritis; Axial Spondyloarthritis; Enthesitis
Keywords: Active psoriatic arthritis; Axial spondyloarthritides; Subcutaneous; Secukinumab in prefilled syringe; Enthesitis; Achilles tendon; AxSpA; PsA
MeSH Terms: conditions — Arthritis, Psoriatic; Axial Spondyloarthritis | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: Randomized Double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AIN457/Secukinumab (Experimental): Secukinumab 150 mg s.c. or Secukinumab 300 mg s.c., respective dose was assigned according to underlying condition, in case of PsA according to severity of concomitant Psoriasis or pre-exposure to anti-TNFα
  Interventions: Biological: Secukinumab
- AIN457/Secukinumab Placebo (Placebo Comparator): Secukinumab Placebo s.c.
  Interventions: Drug: Secukinumab Placebo

INTERVENTIONS:
Biological: Secukinumab — Induction: Week 0,1,2,3 150 mg or 300 mg Secukinumab s.c. Maintenance: 150 mg or 300 mg Secukinumab s.c. every 4 weeks starting at Week 4
  Other Names: AIN457A
  Arms: AIN457/Secukinumab
Drug: Secukinumab Placebo — Induction: Week 0,1,2,3 Secukinumab Placebo s.c. Maintenance: Secukinumab Placebo s.c. every 4 weeks starting at Week 4 until Week 24 followed by 150 or 300 mg Secukinumab s.c. every 4 weeks
  Other Names: AIN457/Secukinumab Placebo
  Arms: AIN457/Secukinumab Placebo

SUMMARY:
The purpose of this study was to demonstrate efficacy, including effects on inflammation by magnetic resonance imaging (MRI) assessments, of secukinumab on Achilles tendon enthesitis for up to 1 year with a primary focus at Week 24, in patients with active Psoriatic Arthritis and axial Spondyloarthritis despite current or previous non-steroidal anti-inflammatory drugs (NSAID) and/or disease modifying anti-rheumatic drug (DMARD) and/or anti-TNFα therapy.

DETAILED DESCRIPTION:
Primary endpoint was at week 24 but there was no interim Clinical Study Report. While Protocol states at chapter 9.7 that a week 24 analysis may be provided (not mandatory as per protocol), all data has been analyzed at week 52.

Some of the secondary endpoints include the whole study period up to week 52 (to address questions on switching placebo to active drug)

ELIGIBILITY:
Key Inclusion Criteria:

- Patients with Psoriatic arthritis: Diagnosis of Psoriatic arthritis as per the Classification criteria for Psoriatic Arthritis (CASPAR criteria) with symptoms for at least 6 months and active Psoriatic arthritis as assessed by ≥ 1 tender joints out of 78 and ≥ 1 swollen joints out of 76 at Baseline (dactylitis of a digit counts as one joint each).

- Patients with Axial Spondyloarthritis: Diagnosis of Axial Spondyloarthritis as per the classification of the Assessment of Spondyloarthritis International Society axial Spondyloarthritis (ASAS) criteria and objective signs of inflammation at Screening (magnetic resonance imaging (MRI) or definite radiographic sacroilitis and/or abnormal C-Reactive Protein) and active disease assessed by total Bath ankylosing spondylitis disease activity index (BASDAI) ≥ 4 (0-10) at Baseline.

* Diagnosis of Achilles tendon enthesitis according to swelling and tenderness at the insertional site of the Achilles tendon into the calcaneus.
* Onset of heel pain ≥ 1 month at Baseline.
* Heel enthesitis that is magnetic resonance imaging (MRI)-positive according to the investigator's judgement.
* Patients who have been exposed to up to two TNFα inhibitors.

Key Exclusion Criteria:

* Chest X-ray or chest magnetic resonance imaging (MRI) with evidence of ongoing infectious or malignant process.
* Previous exposure to secukinumab or other biologic drug directly targeting Interleukin (IL)-17 or Interleukin (IL)-17 receptor.
* Ongoing use of psoriasis treatments / medications (e.g. topical corticosteroids, ultraviolet (UV) therapy) at randomization.
* Patients who have previously been exposed to more than two Tumor necrosis factor (TNF) inhibitors (investigational or approved).
* Patients who have ever received biologic immunomodulating agents (investigational or approved), except those targeting Tumor necrosis factor (TNF) inhibitors.
* Pregnant or nursing (lactating) women.
* History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- Bulgaria (4):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
  - Novartis Investigative Site, Targovishte
- Czechia (4):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Germany (11):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Cottbus
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Wuppertal
- Greece (3):
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Italy (6):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Potenza, PZ
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Bologna
- Novartis Investigative Site, Piešťany, Slovakia
- Spain (11):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Torrelavega, Cantabria
  - Novartis Investigative Site, Mérida, Extremadura
  - Novartis Investigative Site, Ourense, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Cartagena, Murcia
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Pontevedra
- United Kingdom (8):
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Stoke-on-Trent, Staffordshire
  - Novartis Investigative Site, Barnsley
  - Novartis Investigative Site, Cheshire
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Tyne and Wear

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Baraliakos X, Sewerin P, de Miguel E, Pournara E, Kleinmond C, Shekhawat A, Jentzsch C, Wiedon A, Behrens F; ACHILLES study group. Magnetic resonance imaging characteristics in patients with spondyloarthritis and clinical diagnosis of heel enthesitis: post hoc analysis from the phase 3 ACHILLES trial. Arthritis Res Ther. 2022 May 16;24(1):111. doi: 10.1186/s13075-022-02797-8. PMID 35578245
- [Derived] Behrens F, Sewerin P, de Miguel E, Patel Y, Batalov A, Dokoupilova E, Kleinmond C, Pournara E, Shekhawat A, Jentzsch C, Wiedon A, Baraliakos X; ACHILLES study group. Efficacy and safety of secukinumab in patients with spondyloarthritis and enthesitis at the Achilles tendon: results from a phase 3b trial. Rheumatology (Oxford). 2022 Jul 6;61(7):2856-2866. doi: 10.1093/rheumatology/keab784. PMID 34730795
- [Derived] Baraliakos X, Sewerin P, de Miguel E, Pournara E, Kleinmond C, Wiedon A, Behrens F. Achilles tendon enthesitis evaluated by MRI assessments in patients with axial spondyloarthritis and psoriatic arthritis: a report of the methodology of the ACHILLES trial. BMC Musculoskelet Disord. 2020 Nov 21;21(1):767. doi: 10.1186/s12891-020-03775-4. PMID 33220702

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 304 patients were screened. Of these, 94 patients discontinued during screening phase, 6 patients were re-screened and 204 patients completed the screening phase and were randomized in the trial.
Pre-assignment Details: A total of 175 patients (85.8%) completed treatment period 1 (up to Week 24); 29 patients (14.2%) discontinued study treatment in treatment period 1. A total of 170 patients (83.3%) completed treatment period 2 (up to Week 52); 5 patients (2.5%) discontinued in treatment period 2.
Groups:
- Secukinumab: Secukinumab 150 mg or 300 mg s.c., administered at baseline, weeks 1, 2, 3, 4 and every 4 weeks until week 24, followed by Secukinumab 150 or 300 mg s.c. every 4 weeks; respective dose was assigned according to underlying condition, in case of PsA according to severity of concomitant Psoriasis or preexposure to anti-TNFα
- Placebo: Placebo 150 mg or 300 mg s.c., administered at baseline, weeks 1, 2, 3, 4 and every 4 weeks until week 24, followed by Secukinumab 150 or 300 mg s.c. every 4 weeks; respective dose was assigned according to underlying condition, in case of PsA according to severity of concomitant Psoriasis or preexposure to anti-TNFα
Period: Period 1
Arm/Group | Secukinumab | Placebo
Started | 102 | 102
Completed | 91 | 84
Not Completed | 11 | 18
Not completed — Adverse Event | 5 | 3
Not completed — Lack of Efficacy | 3 | 6
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Withdrawal of informed consent | 1 | 5
Period: Period 2
Arm/Group | Secukinumab | Placebo
Started (Completed treatment period 1 and continued to treatment period 2) | 91 | 84
Completed | 89 | 81
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Withdrawal of informed consent | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomized Set: The Randomized set was defined as all patients who were randomized. Unless otherwise specified, mis-randomized patients in the IRT were excluded from the randomized set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Categorical [Count of Participants; unit: Participants] — Number of participants in each age group
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 97 | 95 | 192
    >=65 years | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] — Mean age of participants in each group
  Years | 47.8 (11.33) | 47.7 (11.02) | 47.7 (11.18)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Number of males vs females in Randomized set
  Participants
    Female | 58 | 55 | 113
    Male | 44 | 47 | 91
Race/Ethnicity, Customized [Number; unit: Participants] — Number of participants (Randomized set) by race
  Participants
    Caucasian | 99 | 99 | 198
    Black | 0 | 0 | 0
    Asian | 2 | 1 | 3
    Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number (%) of Patients With Resolution of Achilles Tendon Enthesitis
Description: Number (%) of patients with resolution of Achilles tendon enthesitis (affected foot) as assessed by respective subcomponent of Leeds enthesitis index (LEI) at Week 24.
  The primary analysis was performed via a logistic regression model with the factors treatment, country, and stratification factor diagnosis (PsA or axSpA); patients with a missing assessment were considered as responders if they had already met the response criterion at the time of last assessment.
Time Frame: Week 24
Population: Full analysis set (FAS) included all patients to whom study medication had been assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 102 | 102
Participants | 43 | 32
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; Test type: Superiority; p = 0.136, Regression, Logistic; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.87 to 3.08]

2. Secondary Outcome: Mean Change of Heel Pain
Description: Mean change of heel pain from baseline to Week 24 measured by Numeric Rating Scale (NRS) ranging from 0 to 10, with 0 representing no pain and 10 representing worst pain (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Time Frame: Week 24
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 87 | 85
Scores on a scale | -2.8 (2.99) | -1.9 (2.69)

3. Secondary Outcome: Number (%) of Patients With Improvement of Bone Marrow Edema
Description: Number (%) of patients with an improvement of bone marrow edema from baseline to Week 24 as assessed by the respective subcomponent of the Psoriatic Arthritis Magnetic Resonance Imaging Score (PsAMRIS) in the affected foot.
Time Frame: Week 24
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 44 | 36
Participants | 17 | 12

4. Secondary Outcome: Number (%) of Patients With Resolution of Enthesitis as Assessed by LEI
Description: Number (%) of patients with resolution of enthesitis as assessed by the Leeds enthesitis index (LEI) at Week 24.
Time Frame: Week 24
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 102 | 102
Participants | 31 | 21

5. Secondary Outcome: Mean Change of Physician's Global Assessment of Disease Activity
Description: Mean change of physician's global assessment (PhGA) of disease activity from baseline to Week 24 measured by Visual Analog Scale (VAS) ranging from 0 to 100, with 0 representing not severe and 100 representing very severe.
Time Frame: Week 24
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 88 | 85
mm | -34.88 (25.927) | -18.93 (26.257)

6. Secondary Outcome: Mean Change of Patient's Global Assessment of Disease Activity
Description: Mean change of patient's global assessment (PGA) of disease activity from baseline to Week 24 measured by Visual Analog Scale (VAS) ranging from 0 to 100, with 0 representing not severe and 100 representing very severe.
Time Frame: Week 24
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 82 | 80
mm | -25.87 (31.108) | -16.61 (29.235)

7. Secondary Outcome: Mean Change of Physician's Assessment of Heel Enthesopathy Activity
Description: Mean change of physician's assessment of heel enthesopathy activity from baseline to Week 24 measured by Visual Analog Scale (VAS) ranging from 0 to 100, with 0 representing not severe and 100 representing very severe.
Time Frame: Week 24
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 88 | 85
mm | -38.40 (24.244) | -25.19 (25.250)

8. Secondary Outcome: Mean Change of Patient's Assessment of Heel Enthesopathy Activity
Description: Mean change of patient's assessment of heel enthesopathy activity from baseline to Week 24 measured by Visual Analog Scale (VAS) ranging from 0 to 100, with 0 representing not severe and 100 representing very severe.
Time Frame: Week 24
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 86 | 84
mm | -31.05 (29.135) | -20.77 (30.417)

9. Secondary Outcome: Mean Change in Short Form-36 (SF-36) v2
Description: Mean change in Short Form-36 (SF-36) v2 as an indicator of overall health status
  The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability
Time Frame: Week 24
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 87 | 85
scores on a scale | 8.29 (9.759) | 5.28 (7.285)

10. Secondary Outcome: Percentage of Patients With Resolution of Achilles Tendon Enthesitis After Switching From Placebo to Secukinumab
Description: Percentage of patients with resolution of Achilles tendon enthesitis (affected foot) after switching from placebo to secukinumab at Week 24
Time Frame: Weeks 24 and 52
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 102 | 102
Participants
  Week 24 | 43 | 32
  Week 52 | 66 | 55

11. Secondary Outcome: Mean Change of Heel Pain After Switching From Placebo to Secukinumab
Description: Mean change of heel pain after switching from placebo to secukinumab from Week 24 to week 52 measured by Numeric Rating Scale (NRS) ranging from 0 to 10, with 0 representing no pain and 10 representing worst pain (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Time Frame: Change from week 24 to week 52
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 80 | 79
Scores on a scale | -0.70 (2.291) | -1.43 (2.251)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment at week 52
Description: * Adverse Events (AEs) are any untoward signs or symptoms that occurred during the study treatment.
  * Where a patient reported more than 1 AE with the same preferred term, the AE was counted only once.
  * Where a patient reported more than 1 AE within the same primary system organ class, patient was counted only once at the system organ class level.
Groups:
- Placebo-Secukinumab: Placebo 150 mg or 300 mg s.c., administered at baseline, weeks 1, 2, 3, 4 and every 4 weeks until week 24, followed by Secukinumab 150 or 300 mg s.c. every 4 weeks; respective dose was assigned according to underlying condition, in case of PsA according to severity of concomitant Psoriasis or preexposure to anti-TNFα
Arm/Group | Secukinumab | Placebo-Secukinumab
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/102
Serious Adverse Events (participants affected / at risk) | 7/102 | 6/102
Other Adverse Events (participants affected / at risk) | 33/102 | 34/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=102) | Placebo-Secukinumab (N=102)
Atrial fibrillation (Cardiac disorders) | 1 | 1
Goitre (Endocrine disorders) | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Migraine with aura (Nervous system disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=102) | Placebo-Secukinumab (N=102)
Diarrhoea (Gastrointestinal disorders) | 8 | 5
Nasopharyngitis (Infections and infestations) | 13 | 22
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Headache (Nervous system disorders) | 6 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT02771210/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT02771210/SAP_001.pdf